CLINICAL TRIAL: NCT06770543
Title: Regulatory Post-Marketing Surveillance (rPMS) Study for Leqvio® Pre-filled Syringe(Inclisiran Sodium)
Brief Title: Leqvio rPMS (Regulatory Post-Marketing Surveillance in Korea)
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A1KR01
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Primary Hypercholesterolemia or Mixed Dyslipidemia
Keywords: primary hypercholesterolemia,; mixed dyslipidemia; inclisiran; Leqvio
MeSH Terms: interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inclisiran: Patients who have been treated with inclisiran
  Interventions: Other: Inclisiran

INTERVENTIONS:
Other: Inclisiran — There is no treatment allocation. Patients administered Leqvio by prescription that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Leqvio®

SUMMARY:
This non-interventional study is a mandatory regular Post Marketing Surveillance(rPMS) granted by the Korean health authorities, and is conducted to assess the effectiveness and safety of Leqvio® Pre-filled Syringe(inclisiran sodium) in routine clinical practice for the approved indications (primary hypercholesterolemia or mixed dyslipidemia).

ELIGIBILITY:
Inclusion Criteria:

If a subject meets all of the following criteria, he/she can participate in this study:

1. Adult patients(18 years or older) who have hypercholesterolemia or mixed dyslipidemia and are prescribed Leqvio® Pre-filled Syringe(inclisiran sodium) according to domestically approved product information in real clinical practice
2. Patients who are unable to reach LDL-C target with maximum tolerated dose of statin, or patients with statin intolerance
3. Patients who provided consent to participate in the study(informed consent form)

Exclusion Criteria:

A subjects who meets any of the following criteria cannot participate in this study:

1. Contraindications in accordance with domestic prescribing information
2. Patients participating in clinical trials of other investigational drugs
3. Patients who do not provide consent to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve patients who received at least one dose of Leqvio for the treatment of primary hypercholesterolemia or mixed dyslipidemia according to the current label information in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2031-01-02 (Estimated); Study Completion 2031-01-02 (Estimated)

PRIMARY OUTCOMES:
Incidences of adverse events/adverse drug reactions (AEs/ADRs) | up to 15 months
  Cumulative incidences of AEs, ADRs, SAEs, Serious ADR(SADRs), Unexpected AEs, and Unexpected ADRs due to Leqvio® Pre-filled Syringe(inclisiran sodium) during the observation period ["The term "unexpected" means that it is not listed in the domestic labeling(according to health authority regulations)]

SECONDARY OUTCOMES:
Change from baseline in low-density lipoprotein-cholesterol (LDL-C) and lipid profiles | Baseline, Months 3, 9 and 15
  Effectiveness of Leqvio® Pre-filled Syringe (inclisiran sodium) through changes in LDL-C and lipid profiles (total cholesterol, Apolipoprotein B (ApoB), non high-density lipoprotein cholesterol (non-HDL-C), Apolipoprotein A-1 (ApoA1), High Density Lipoprotein Cholesterol (HDL-C), Lipoprotein(a) (Lp(a)) and triglyceride).
Impact of subjects' baseline characteristics and medication usage on cumulative incidence of AEs and SAEs | up to 15months
  Impact of subjects' baseline characteristics(age, gender, pregnancy, BMI, lipid profile, cardiovascular risk factors and comorbidities) and medication & non-medication(reason for using the drug, usage period, amount of use, concomitant medications) on cumulative incidence of AEs and SAEs during the observation period.
Impact of subjects' baseline characteristics and medication usage on changes from baseline in LDL-C and lipid profiles | up to 15 months
  Impact of subjects' baseline characteristics(age, gender, pregnancy, BMI, lipid profile, cardiovascular risk factors and comorbidities) and medication & non-medication(reason for using the drug, usage period, amount of use, concomitant medications) on the changes in LDL-C and lipid profiles after treatment compared to baseline.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu

IPD SHARING:
Plan to Share IPD: No